CLINICAL TRIAL: NCT06377540
Title: MT2022-60: A Phase II Study of Pembrolizumab+ BEAM Conditioning Regimen Before Autologous Stem Cell Transplant (ASCT) Followed by Pembrolizumab Maintenance in Patients of Relapsed or Refractory Classic Hodgkin Lymphoma
Brief Title: MT2022-60: Ph 2 Study of Pembro+ BEAM With ASCT for Relapsed Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022LS174
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Autologous Stem Cell Transplant; Classic Hodgkin Lymphoma
Keywords: BEAM; cHL; ASCT
MeSH Terms: interventions — pembrolizumab; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab+BEAM followed by ASCT followed by Pembrolizumab maintenance for 1 year. (Experimental): Patients will receive Pembrolizumab before BEAM ASCT followed by Pembrolizumab maintenance for 1 year. Patients will receive 200 mg Pembrolizumab starting at day - 28 before stem cell transplant until 1 year after autologous stem cell transplant.
  Interventions: Drug: Pembrolizumab; Procedure: Autologous stem cell transplant; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan

INTERVENTIONS:
Drug: Pembrolizumab — Patients will receive 200 mg Pembrolizumab on Day -28 and Day -6 by IV infusion.
  Pembrolizumab 200 mg IV will resume at day 30+ after ASCT every 3 weeks for 1 year.
  Other Names: Keytruda; MK-3475
Procedure: Autologous stem cell transplant — On day 0 the stem cells will be infused immediately after thawing over 15-60 minutes per institutional guidelines.
  Other Names: ASCT
Drug: Carmustine — Patient will receive a single dose of BCNU on day -6, dose of 300 mg/m2 by IV infusion.
  Other Names: BCNU; BICNU
Drug: Etoposide — Etoposide will be given at dose 100 mg/m2 BID intravenously on days -5, - 4, -3, and -2.
Drug: Cytarabine — Cytarabine will be given at dose 100 mg/m2 BID intravenously on days -5, -4, - 3, and -2.
  Other Names: Ara-C
Drug: Melphalan — Melphalan will be given at dose of 140 mg/m2 intravenously on day -1 in a single 20 minute infusion; dose will be based on actual body weight but capped at 3.6 mg/kg as part of BEAM conditioning.

SUMMARY:
This is a Phase 2 single arm study to evaluate efficacy and safety of Pembrolizumab before with BEAM ASCT followed by Pembrolizumab maintenance for 1 year. Patients will receive 200 mg Pembrolizumab Q3week starting at day - 28 before stem cell transplant until 1 year after autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for autologous stem cell transplant (ASCT) with BEAM conditioning regimen
* KPS greater than 70 or ECOG ≤ 1
* Adequate organ function and blood counts within 14 days of study registration
* Participants who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization.
* Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening.
* HIV-infected participants must have well-controlled HIV on ART

Exclusion Criteria:

* Patients with prior history of any grade 2 or higher autoimmune reaction to PD-1 inhibitors, necessitating permanent discontinuation of the PD-1 inhibitor or necessitating systemic immunosuppressants.
* Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Has received any chemotherapy within 3 weeks prior to the first dose of study intervention
* Has known active CNS disease.
* History of or active autoimmune disease, or other syndrome that requires systemic steroids or autoimmune agents. Exceptions: Participants with vitiligo, resolved childhood asthma or atopy, hypothyroidism, or Sjogren's syndrome, as well as participants requiring only intranasal steroids, intermittent use of bronchodilators, local steroid injections, or physiologic replacement doses of prednisone (≤ 10 mg/d) may enroll.
* Has had an allogenic tissue/solid organ transplant.
* Pregnant or breastfeeding as agents used in this study are Pregnancy Category D (positive evidence of risk). Females of childbearing potential must have a negative pregnancy test (serum or urine) within 14 days of study registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Baseline to 1 year post-ASCT
  Number of participants with progression free survival at 1 year post transplant.
  Time from date of study enrollment to date of first documented progression, or death. Patients who do not progress or die at the time of analysis will be censored at their last known date alive.

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline to 2 years post-ASCT
  Time from date of study enrollment to date of death. Patients who do not die at the time of analysis will be censored at their last known date alive.
Progression-free survival (PFS) | Baseline to 2 years post-ASCT
  Number of participants with progression free survival at 1 year post transplant.
  Time from date of study enrollment to date of first documented progression, or death. Patients who do not progress or die at the time of analysis will be censored at their last known date alive.
Non-relapse mortality (NRM) | Day 100 post-ASCT
  Number of participants experiencing death without relapse.
Overall Survival (OS) | Baseline to 5 year post-ASCT
  Time from date of study enrollment to date of death. Patients who do not die at the time of analysis will be censored at their last known date alive.
Complete Radiologic Response Rate | Day 28
  Participants experiencing complete radiologic response rate at day 28 post-ASCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No